CLINICAL TRIAL: NCT06095154
Title: CTV Delineation Based Solely on Geometric Expansion From GTV in Nasopharyngeal Carcinoma: A Prospective, Multi-center, Randomized Controlled Phase III Clinical Study
Brief Title: CTV Delineation Based Solely on Geometric Expansion From GTV in Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC009
Record Dates: First submitted 2023-10-14; First posted 2023-10-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Carcinoma by AJCC V8 Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): GTVp (70Gy/33Fx): Gross tumor as seen on imaging and nasopharyngoscopy. CTVp1 (60Gy/33Fx): None. CTVp2 (54Gy/33Fx): GTVp + 10 mm + entire nasopharyngeal mucosa. GTVn: Lymph nodes as seen on imaging. CTVn: Defined according to CACA/CMDA guidelines.
  Interventions: Radiation: CTV Delineation Based on Geometric Expansion From GTV in Nasopharyngeal Carcinoma
- Control Group (No Intervention): GTVp (70Gy/33Fx): Gross tumor as seen on imaging and nasopharyngoscopy. CTVp1 (60Gy/33Fx): GTVp + 5 mm + entire nasopharyngeal mucosa. CTVp2 (54Gy/33Fx): GTVp + 10 mm + high-risk anatomical structures. GTVn: Lymph nodes as seen on imaging. CTVn: Defined according to CACA/CMDA guidelines.

INTERVENTIONS:
Radiation: CTV Delineation Based on Geometric Expansion From GTV in Nasopharyngeal Carcinoma — CTVp2 is generated by expanding GTVp by 10 mm and including the nasopharyngeal mucosa.
  Arms: Experimental Group

SUMMARY:
This is a randomized, phase III, prospective, multi-center trial in newly diagnosed nasopharyngeal carcinoma (NPC) patients without distant metastasis. The aim of this study is to evaluate the efficacy and safety of modified IMRT, of which CTV delineation was only based on geometric expansion from GTV.

DETAILED DESCRIPTION:
All enrolled patients underwent intensity-modulated radiation therapy (IMRT). The IMRT technique was selected based on the equipment available at each treatment center and the patients' preferences, including IMRT, VMAT, or TOMOTHERAPY. According to our study design, all enrolled patients will be randomly assigned in a 1:1 ratio before radiation therapy. The target area definitions are based on the international ICRU reports No. 50 and No. 60. The specific target area definitions and prescribed doses for the two groups are as follows:

1. GTVp (70Gy/33Fx) Experimental Group: Gross tumor as seen on imaging and nasopharyngoscopy; Control Group: Gross tumor as seen on imaging and nasopharyngoscopy.
2. CTVp1 (60Gy/33Fx) Experimental Group: None; Control Group: GTVp + 5 mm + entire nasopharyngeal mucosa.
3. CTVp2 (54Gy/33Fx) Experimental Group: GTVp + 10 mm + entire nasopharyngeal mucosa; Control Group: GTVp + 10 mm + high-risk anatomical structures.
4. GTVn Experimental Group: Lymph nodes as seen on imaging; Control Group: Lymph nodes as seen on imaging.
5. CTVn Experimental Group: Defined according to CACA/CMDA guidelines; Control Group: Defined according to CACA/CMDA guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis (pathologically confirmed by nasopharyngeal biopsy) was nasopharyngeal carcinoma;
2. No distant metastatic;
3. Patients with baseline MRI date of nasopharynx and neck, and completed the first course of treatment in our hospital;
4. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1;
5. Signing informed consent;
6. Follow up regularly and comply with test requirements.

Exclusion Criteria:

1. Disease progression during IMRT;
2. Previous malignancy or other concomitant malignant diseases;
3. The evaluation information of tumor efficacy can not be obtained;
4. Receive blind treatment in other clinical research;
5. Have or are suffering from other malignant tumors within 5 years (except non- melanoma skin cancer or pre-invasive cervical cancer);
6. Serious complications, such as uncontrolled hypertension, coronary heart disease, diabetes, heart failure, etc;
7. Active systemic infection;
8. No or limited capacity for civil conduct;
9. The patient has a physical or mental disorder, and the researcher considers that the patient is unable to fully or fully understand the possible complications of this study;
10. Pregnancy or lactation period;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Local failure-free survival (LFFS) | 3 years
  The duration of time to LFFS was calculated from the date of histological diagnosis until documented treatment local failure or death from any cause.

SECONDARY OUTCOMES:
overall survival | 3 years
  time from the date of the start of chemotherapy to death due to any cause
Regional failure-free survival | 3 years
  The regional relapse-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to the date of nodal relapse or death from any cause, whichever occurred first. Their differences will be compared between treatment arms using the log-rank test.
Distant metastasis-free survival | 3 years
  The distant metastasis-free survival rate will be estimated using Kaplan-Meier
Patient's quality-of-life | 3 years
  uropean Organization for Research and Treatment of Cancer Quality-of-Life Head

CONTACTS AND LOCATIONS:
Overall Officials: Shaojun Lin, DR, Study Chair — Fujian Cancer Hospital
Locations (1):
- Fujian Cancer hospital, Fuzhou, Fujian, China